CLINICAL TRIAL: NCT01852864
Title: A Study of the Early Biological Effects of Testosterone Suppression in Prostate Cancer Using Neoadjuvant Degarelix Prior to Radical Prostatectomy
Brief Title: Degarelix Before Radical Prostatectomy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cambridge (Other)
Responsible Party: Principal Investigator, Greg Shaw, Clinical Lecturer in Urology, University of Cambridge
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11/H0311/2
Record Dates: First submitted 2013-05-06; First posted 2013-05-14 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; testosterone; castration; degarelix; proliferation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Degarelix treated group (Experimental): 240mg degarelix s.c. injection to be administered 7 days prior to radical prostatectomy for high/intermediate risk prostate cancer.
  Interventions: Drug: 240mg degarelix s.c. injection

INTERVENTIONS:
Drug: 240mg degarelix s.c. injection — 7 days prior to radical prostatectomy the patient will have a subcutaneous injection of 240mg degarelix.
  Other Names: medical castration

SUMMARY:
The biological effects of castration on prostate cancers will be studies by administration of degarelix prior to radical prostatectomy.

The effects will be studied by analysis of gene expression and immunohistochemistry focusing on markers of proliferation and apoptosis of samples taken at the time of radical prostatectomy (7 days after administration of degarelix).

Tumours from patients treated with neo-adjuvant degarelix will be compared with tumours from patients who have not been medically castrated.

ELIGIBILITY:
Inclusion Criteria:

* Intermediate/high risk prostate cancer
* Patient eligible for and wanting surgery

Exclusion Criteria:

* Inability to consent
* Previous thromboembolism/arrhythmias
* contraindication to degarelix or surgery

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
proliferative index defined by immunohistochemistry for ki67 | at surgery, 7 days after administration of degarelix

SECONDARY OUTCOMES:
Gene expression levels measured by microarray | At surgery 7 days after degarelix administration

CONTACTS AND LOCATIONS:
Overall Officials: David Neal, BSc MS FRCS, Study Chair — Cambridge University
Locations (1):
- Cambridge University Hopital NHS Trust, Cambridge, Cambridgeshire, United Kingdom